CLINICAL TRIAL: NCT05161091
Title: Efficacy of Orosol® in the Treatment of Chemo- and Radiation-induced Mucositis. Randomized, Double-blind, Placebo-controlled Trial.
Brief Title: Efficacy of Orosol® in the Treatment of Chemo- and Radiation-induced Mucositis.
Acronym: OROSOL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RBHP 2021 DEVOIZE (OROSOL); 2021-A00488-33 (Other: 2021-A00488-33)
Record Dates: First submitted 2021-11-22; First posted 2021-12-16 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Oral Mucositis
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Radio-induced oral mucositis / Medical Device (Experimental): Patient with radio-induced oral mucositis at least grade 2 treated with experimental medical device
  Interventions: Device: Topical application of Orosol®
- Radio-induced oral mucositis / Placebo comparator (Placebo Comparator): Patient with radio-induced oral mucositis at least grade 2 treated with placebo
  Interventions: Device: Topical application of Placebo comparator
- Chemo-induced oral mucositis / Medical Device (Experimental): Patient with chemo-induced oral mucositis at least grade 2 treated with experimental medical device
  Interventions: Device: Topical application of Orosol®
- Chemo-induced oral mucositis / placebo comparator (Placebo Comparator): Patient with chemo-induced oral mucositis at least grade 2 treated with placebo
  Interventions: Device: Topical application of Placebo comparator

INTERVENTIONS:
Device: Topical application of Orosol® — Orosol® is a 20 ml aluminum bottle equipped with a spray without propellant gas for local application. Simply shake the bottle gently, apply the product to the injured surface by pressing your finger on the spray to deliver the product (4 to 5 times so as to form a thin film on the surface of the mouth) . It is recommended to use Orosol® every 2 hours at the start of treatment and then 3 to 4 times a day. The maximum duration of treatment will be 28 days. Eating or drinking should be avoided for the first 15 to 30 minutes after applying the product.
  Arms: Chemo-induced oral mucositis / Medical Device; Radio-induced oral mucositis / Medical Device
Device: Topical application of Placebo comparator — Placebo comparator is a 20 ml aluminum bottle equipped with a spray without propellant gas for local application. Simply shake the bottle gently, apply the product to the injured surface by pressing your finger on the spray to deliver the product (4 to 5 times so as to form a thin film on the surface of the mouth) . It is recommended to use Placebo comparator every 2 hours at the start of treatment and then 3 to 4 times a day. The maximum duration of treatment will be 28 days. Eating or drinking should be avoided for the first 15 to 30 minutes after applying the product.
  Arms: Chemo-induced oral mucositis / placebo comparator; Radio-induced oral mucositis / Placebo comparator

SUMMARY:
Oral mucositis is one of the most debilitating side effects of radiation therapy and various forms of chemotherapy, especially for head and neck cancers and hematopoietic stem cell transplants.

It is a consequence of the cytostatic effects of anticancer treatments on rapidly renewing cells of the oral mucosa; An ulcer appears which will increase in size due to subsequent bacterial, fungal and / or viral growth, while the leakage of toxins through damaged capillaries causes irritation and a burning sensation. Proteolytic enzymes, known to destroy the extracellular matrix, inhibit cell regeneration and healing.

Depending on the severity of the ulceration, infection and feeding possibilities, mucositis is scored between grade 0 (absent) and grade 4 (maximum) (according to the WHO (World Health Organization) classification or the NCI-CTCAE (National Cancer Institute-Common Terminology Criteria for Adverse Events), the latter degree most often requiring a modification of the anticancer treatment which may have an impact on the prognosis of the disease.

Although, theoretically, mucositis is easy to treat because it only requires simple cleaning of the ulcers and stimulation of the growth of the underlying healthy cells to make up for the loss of substance, there are currently only limited symptomatic treatments available.

DETAILED DESCRIPTION:
Oral mucositis is one of the frequent and disabling effects of radiotherapy and chemotherapy, with an impact on the quality of life of patients and induced or prolonged hospital stays. It is a consequence of the cytostatic effects of anticancer treatments on rapidly renewing cells of the oral mucosa. Proteolytic enzymes, known to destroy the extracellular matrix, inhibit cell regeneration and healing. Treatment is currently symptomatic, with little effectiveness. Orosol® is a medical device, osmotically active viscous solution. Applied to the surface of an ulcer, it forms a film and mechanically attracts the hypotonic fluid present under the injured surface, thus cleaning the ulcer of all contaminants present on the surface (dead cells, cell debris, bacterial toxins and chemical agents. toxic) and reducing pain and burning sensation. This mechanical action also cleanses the ulcer of toxic substances that inhibit cell growth and paves the way for healing. This device (class 1) is a medical device that complies with the requirements set by European regulations for the treatment of oral mucositis and has shown improvement in a preliminary study in patients with chemo-induced mucositis. However, its effectiveness has not yet been tested in the case of radiation-induced mucositis. The main objective of the research is to demonstrate the effectiveness of the curative treatment with Orosol® on the symptoms of chemo-induced or radiation-induced mucositis in patients treated for cancer by the evaluation at 28 days of the evolution of the mucositis via mucositis (WHO and NCI-CTCAE v3.0 scales) and food (WHO scales and functional signs of NCI-CTCAE v4.0) scores. The secondary objectives consist in evaluating during the treatment the mucositis score, the general state of health of the mouth, the burning sensation, the intensity of the pain on D1, D3, D5, D7, D14, D21 and D28 as well as analgesic consumption, the incidence of new ulcers, changes in anti-cancer treatment linked to mucositis and the tolerance of the treatment.

This is a prospective, randomized, double-blind, bicenter study to establish CE compliance in a new indication. 54 adult patients, treated by chemotherapy for haematological cancer or radiotherapy or radio-chemotherapy for head and neck cancer, with CTCAE grade ≥ 2 mucositis and agreeing not to take any treatment other than that studied (except the treatment symptomatic of mucositis recommended by the WHO), will be recruited during their treatment in the specialized services of the Clermont-Ferrand University Hospital or the Jean Perrin Center over a period estimated at 24 months. After information, collection of consent and verification of the selection criteria, patients will receive according to randomization (1: 1 stratified according to radio / chemotherapy) either the active treatment or a placebo. During the first visit, a clinical examination with evaluation of the grade of mucositis (WHO scale and clinical signs NCI-CTCAE v3.0), photographs of ulcers (retrospective control), evaluation of the state of the mouth (OAG (Oral Assessment Guide) grid), difficulty in feeding by the oral route (functional signs NCI- CTCAE v4.0) will be performed as well as assessments (VAS (Visual Analogic Scales) of pain and burning sensations before and 30 minutes after treatment. Visits are scheduled on D3, D5, D7, D14, D21 and D28 with clinical examination, photographs, evaluations of the condition of the mouth, difficulty in feeding, pain and burning sensation, collection of any adverse effects and changes in the anti-cancer treatment if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, male or female, either

  * treated with chemotherapy for hematological cancer (leukemia, lymphoma) and suffering from grade 2 to 4 mucositis (according to WHO / NCI-CTCAE), or
  * treated with radiotherapy or radio-chemotherapy (cisplatin or cetuximab) for head and neck cancer and suffering from grade 2 to 4 mucositis (according to WHO / NCI-CTCAE),
* Agreeing not to take any treatment for mucositis other than the treatment proposed in this study, apart from the classic symptomatic treatment for mucositis recommended by WHO.
* Able to give informed consent to participate in research.
* Beneficiary of a Social Security scheme.

Exclusion Criteria:

* A woman who is pregnant, breastfeeding, or may be.
* Major subject under guardianship, curators, deprived of liberty, or under the safeguard of justice.
* Medical and / or surgical history deemed by the investigator to be incompatible with the study because it would invalidate any reliable assessment.
* General state of health considered pejorative (Karnofsky index <60).
* Type 1 or type 2 diabetic subject (presence of honey in Orosol®).
* Subject on an anticoagulant (AVK or AOD) (interaction of the cranberry contained in Orosol® with anticoagulants (in particular warfarin) with instability of the International Normalized Ratio; the AODs can potentially present the same type of interaction).
* History of administration of the treatment (or equivalent) in the study.
* Anticipated difficulties in reading / understanding the protocol and its questionnaires.
* Subjects in the exclusion period from another clinical trial
* Refusal of participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the effectiveness of the curative treatment with Orosol® on mucositis score (WHO) | At day 28
  Evolution the symptoms of chemo-induced or radiation-induced mucositis by collecting the mucositis score according to the World Health Organization scale (from 0 (absence of mucositis) to 4 (Oral feeding not possible, enteral (tube) or parenteral feeding indicated))
Demonstrate the effectiveness of the curative treatment with Orosol® on mucositis score (NCI-CTCAE v3.0) | At day 28
  Evolution the symptoms of chemo-induced or radiation-induced mucositis by collecting the mucositis score according to the National Cancer Institute Common Terminology Criteria for Adverse Events (clinical scale) (v 3.0) (from 0 (absence of mucositis) to 4 (Necrosis, spontaneous hemorrhage))
Demonstrate the effectiveness of the curative treatment with Orosol® on oral feeding (NCI-CTCAE v4.0) | At day 28
  Evolution the symptoms of chemo-induced or radiation-induced mucositis by collecting the difficulty in feeding orally with the functional signs scale from the National Cancer Institute Common Terminology Criteria for Adverse Events (functional scale) (v 4.0) (from 0 (absence of mucositis) to 4 (Necrosis, Vital prognosis engaged))

SECONDARY OUTCOMES:
Assessment of general state of health of the mouth with Oral Assessment Guide (OAG) scale "item voice" | At day 1, 3 , 5, 7, 14, 21 and 28
  The OAG "item voice" scale is a scale from 1 (Normal) to 3 (highly impacted) assessing the difficulty of speaking
Assessment of general state of health of the mouth with Oral Assessment Guide (OAG) scale "item swallowing" | At day 1, 3 , 5, 7, 14, 21 and 28
  The OAG "item swallowing" scale is a scale from 1 (Normal) to 3 (highly impacted) assessing the difficulty of swallowing
Assessment of general state of health of the mouth with Oral Assessment Guide (OAG) scale "item tongue aspect" | At day 1, 3 , 5, 7, 14, 21 and 28
  The OAG "item tongue aspect" scale is a scale from 1 (pink, wet and presence of taste buds) to 3 (cracked, blistered) assessing the aspect of the tongue
Assessment of general state of health of the mouth with Oral Assessment Guide (OAG) scale "item salivation" | At day 1, 3 , 5, 7, 14, 21 and 28
  The OAG "item salivation" scale is a scale from 1 (normal) to 3 (absence of salivation) assessing the hyposialia
Assessment of general state of health of the mouth with Oral Assessment Guide (OAG) scale "item mucous membrane and gums" | At day 1, 3 , 5, 7, 14, 21 and 28
  The OAG "item mucous membrane and gums" scale is a scale from 1 (pink and wet) to 3 (ulcerations and / or bleeding) assessing the state of aggression of the mucous membranes
Assessment of general state of health of the mouth with Oral Assessment Guide (OAG) scale "teeth" | At day 1, 3 , 5, 7, 14, 21 and 28
  The OAG "item teeth" scale is a scale from 1 (clean and free of debris) to 3 (widespread plaques and debris on all damaged gums and teeth) assessing the state of aggression of the teeth
Assessment of general state of health of the mouth with Oral Assessment Guide (OAG) scale "lips" | At day 1, 3 , 5, 7, 14, 21 and 28
  The OAG "item lips" scale is a scale from 1 (smooth, dewy and damp) to 3 (ulcerations or bleeding) assessing the state of aggression of the lips
Burning sensation | At day 1, 3 , 5, 7, 14, 21 and 28
  Assessment of burning symptom with visual analogical scale (from 0 (absence of burning sensation to 10 (strongest burning sensation imaginable)
Pain intensity | At day 1, 3 , 5, 7, 14, 21 and 28
  Assessment of pain with visual analogical scale (from 0 (absence of pain sensation to 10 (strongest pain sensation imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Devoize, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - Centre Jean-Perrin, Clermont-Ferrand
  - CHU clermont-ferrand, Clermont-Ferrand

REFERENCES:
- [Background] Feller L, Essop R, Wood NH, Khammissa RA, Chikte UM, Meyerov R, Lemmer J. Chemotherapy- and radiotherapy-induced oral mucositis: pathobiology, epidemiology and management. SADJ. 2010 Sep;65(8):372-4. PMID 21133051
- [Background] Velez I, Tamara LA, Mintz S. Management of oral mucositis induced by chemotherapy and radiotherapy: an update. Quintessence Int. 2004 Feb;35(2):129-36. PMID 15000636
- [Background] Peterson DE. New strategies for management of oral mucositis in cancer patients. J Support Oncol. 2006 Feb;4(2 Suppl 1):9-13. PMID 16499139